CLINICAL TRIAL: NCT01836991
Title: Phase 2 Study of D2 and D2+ Radical Surgery for the Treatment of Advanced Distal Gastric Cancer
Brief Title: D2 and D2+ Radical Surgery for the Treatment of Advanced Distal Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS-ADGC
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; surgery; surgery safety; effect
MeSH Terms: conditions — Stomach Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D2 surgery (Other): D2 surgery(No.1、No.3、No.4sb、No.4d、No.5、No.6、No.7 and No.8a、No.9、No.11p、No.12a lymph node)
  Interventions: Procedure: surgery
- D2+ surgery (Experimental): D2+ surgery(D2+8p、12b、13、14v lymph node)
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery

SUMMARY:
The purpose of this study is to evaluate the safety and the effect of D2 and D2+ radical surgery for the treatment of advanced distal gastric cancer.

DETAILED DESCRIPTION:
To evaluate the safety and the disease-free survival time(DFS) and overall survival time(OS) of D2 and D2+ radical surgery for the treatment of advanced distal gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18 to 70 years old.
* The preoperative evaluation: distal gastric cancer patients, ≥ T2 or N +; or staging II, IIIA, IIIB.
* Karnofsky score ≥ 70, life expectancy > 6 months.
* Endoscopic biopsy diagnosis of gastric cancer, excluding non-Hodgkin's lymphoma, leiomyosarcoma and other mesenchymal tumors.
* the blood and biochemical indicators of the subjects must meet the following criteria: Hb ≥ 9 g / dl; WBC ≥ 4,000 / mm3, ≤ 12000 / mm3; PLT ≥ 100,000/mm3;
* GOT, GPT within twice the institutional limit,serum total bilirubin < 1.5 times the upper limit of normal, serum creatinine< 1.25 times the upper limit of normal
* have not received prior chemotherapy, radiotherapy and biological therapy. signed informed consent.
* must accept the standard D2 or D2 + radical gastrectomy.
* with good compliance.

Exclusion Criteria:

* pregnancy, breast-feeding women.
* allergy with chemotherapy drugs or metabolic disorder.
* the history of organ transplants (including bone marrow transplantation and autologous peripheral stem cell transplantation).
* had long received systemic steroid treatment (Note: short-term users of withdrawal > 2 weeks can be selected.)
* The existence of the peripheral nervous system disorders or significant neurological disorders and a history of central nervous system disorders.
* patients with severe infection requires treatment.
* patients associated with dysphagia, active peptic ulcer, incompleteness intestinal obstruction, active gastrointestinal bleeding, perforation.

severe liver disease (such as cirrhosis), kidney disease, respiratory disease or uncontrollable diabetes.

* with other malignancies which were not cured.
* EKG abnormalities or heart disease with apparent clinical symptoms, including congestive heart failure, coronary heart disease with symptoms, uncontrollable arrhythmia, hypertension, and heart attack within 12 months or III or IV grade myocardial infarction. Coronary heart disease with symptoms, uncontrollable arrhythmia, hypertension, and heart attack within 12 months or III or IV grade myocardial infarction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
the disease-free survival time | 3 years
the overall survival time | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: xiangdong Cheng, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Xu ZY, Hu C, Chen S, Du YA, Huang L, Yu PF, Wang LJ, Cheng XD. Evaluation of D2-plus radical resection for gastric cancer with pyloric invasion. BMC Surg. 2019 Nov 20;19(1):172. doi: 10.1186/s12893-019-0605-6. PMID 31747885
- [Derived] Yu P, Du Y, Xu Z, Huang L, Cheng X. Comparison of D2 and D2 plus radical surgery for advanced distal gastric cancer: a randomized controlled study. World J Surg Oncol. 2019 Feb 6;17(1):28. doi: 10.1186/s12957-019-1572-1. PMID 30728027